CLINICAL TRIAL: NCT01751750
Title: Grape Polyphenol Kinetics in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Janet Novotny (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Janet Novotny, Principal Investigator, USDA Beltsville Human Nutrition Research Center
Organization: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HS38
Record Dates: First submitted 2012-12-10; First posted 2012-12-18 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — whole grape extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Grape (Other)
  Interventions: Other: Grape

INTERVENTIONS:
Other: Grape — 16 oz. of Concord grape juice (8 oz. consumed 2 times per day; total dose of approximately 1.2 g phenolic compounds per day), 250 mg resveratrol provided as a capsule (commercially available supplement; 125 mg consumed 2 times per day), and 1 g grape seed polyphenol extract provided as a capsule (commercially available supplement; 0.5 g consumed 2 times per day).

SUMMARY:
The objectives of this study are the following: 1) to confirm that the administration of grape juice, resveratrol, and grape seed polyphenol extract results in a similar plasma and urinary metabolic profile in aged humans compared to rats, 2) to confirm that a combined administration of grape juice, resveratrol, and grape seed polyphenol extract result in a similar plasma and urinary metabolic profile in adults with tendencies toward metabolic syndrome compared to non-obese healthy humans, and 3) to identify the anti-inflammatory effects of the combined administration of grape juice, resveratrol, and grape seed polyphenol extract.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Age <60 years at beginning of study
* Fasting glucose > 126 mg/dl
* Blood pressure > 160/100
* Fasting total blood cholesterol > 280 mg/dl
* Fasting triglycerides > 300 mg/dl
* Presence of kidney disease, liver disease, gout, hyperthyroidism, untreated or unstable hypothyroidism, certain cancers, gastrointestinal disease, pancreatic disease, other metabolic diseases, or malabsorption syndromes
* Presence of type 2 diabetes requiring the use of oral antidiabetic agents or insulin
* History of bariatric or certain other surgeries related to weight control
* Smokers or other tobacco users (during 6 months prior to the start of the study)
* Consumption of more than 3 servings of tea, wine, or grape juice per day
* Use of supplements containing grape extracts or products
* Use of antibiotics during the intervention or for 3 weeks prior to the intervention period
* History of eating disorders, dietary patterns, or supplement use which will interfere with the goal of the intervention
* Volunteers who have lost 10% of body weight within the last 4 months
* Volunteers who are unable or unwilling to give informed consent or communicate with study staff
* Volunteers who self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Max Age: 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Plasma polyphenols | 6 hours
  Blood will be analyzed for polyphenols and polyphenol metabolites.
Urinary polyphenols | 6 hours
  Urine will be analyzed for polyphenols and polyphenol metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Novotny, Ph.D., Principal Investigator — USDA Beltsville Human Nutrition Research Center
Locations (1):
- USDA Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Novotny JA, Chen TY, Terekhov AI, Gebauer SK, Baer DJ, Ho L, Pasinetti GM, Ferruzzi MG. The effect of obesity and repeated exposure on pharmacokinetic response to grape polyphenols in humans. Mol Nutr Food Res. 2017 Nov;61(11):10.1002/mnfr.201700043. doi: 10.1002/mnfr.201700043. Epub 2017 Aug 29. PMID 28654207